CLINICAL TRIAL: NCT05594290
Title: Window-of-opportunity Study of Chemo-immunotherapy in Patients With Resectable Merkel Cell Carcinoma Prior to Surgery: the MERCURY Trial
Brief Title: Chemo-immunotherapy in Patients With Resectable Merkel Cell Carcinoma Prior to Surgery
Acronym: MERCURY
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gruppo Oncologico del Nord-Ovest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MERCURY
Record Dates: First submitted 2022-10-17; First posted 2022-10-26 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Merkel Cell Carcinoma
Keywords: Merkel Cell Carcinoma; Chemo-immunotherapy; Retifanlimab; Surgery
MeSH Terms: conditions — Carcinoma, Merkel Cell | interventions — Cisplatin; Etoposide

STUDY DESIGN:
Intervention Model Description: Phase 2, multicentre, single-arm, open-label clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Preoperative arm (Experimental): Patients will be treated with one cycle of chemo-immunotherapy with retifanlimab (500 mg day 1), cisplatin (25 mg/sqm i.v. day 1, 2 ) or carboplatin (AUC 4 i.v., day 1 - in patients unsuited or unfit for cisplatin) and etoposide (100 mg/sqm iv. day 1, 2, 3).
  After receiving the short-course preoperative chemo-immunotherapy study regimen, patients will undergo standard radical surgery. After surgery, patients will receive adjuvant radiation therapy if indicated
  Interventions: Drug: Retifanlimab; Drug: Cisplatin; Drug: Etoposide

INTERVENTIONS:
Drug: Retifanlimab — Retifanlimab i.v. 500 mg day 1
Drug: Cisplatin — Cisplatin 25 mg/sqm i.v. day 1, 2 (recommended platinum agent) or carboplatin AUC 4 i.v., day 1 (in patients unsuited or unfit for cisplatin)
Drug: Etoposide — Etoposide 100 mg/sqm iv. day 1, 2, 3

SUMMARY:
This is a window-of-opportunity study for patients with resectable Merkel Cell Carcinoma.

The aim of this study is to test the activity of a course of chemo-immunotherapy followed by surgery in patients with operable Merkel cell carcinoma.

Participants will receive one cycle of retifanlimab plus platinum-etoposide chemotherapy prior to their scheduled surgery.

DETAILED DESCRIPTION:
This is a multicenter, single-arm, open-label, phase 2 Window-of-opportunity trial to assess the activity of 1 cycle of preoperative retifanlimab plus platinum-etoposide chemo-immunotherapy regimen in patients with resectable MCC (stage IIA-III).

Patients who meet the eligibility criteria will be treated with one cycle of chemo-immunotherapy.

After receiving the short-course preoperative chemo-immunotherapy study regimen, patients will undergo standard radical surgery between weeks 5 and 6 from enrollment. After surgery, patients will receive adjuvant radiation therapy, if indicated, and afterwards, standard follow up will be started as per clinical practice and guidelines.

Baseline radiological assessments will include chest/abdomen/pelvis CT scan with contrast and CT scan of additional anatomical sites should be performed if the primary tumor is elsewhere.

The enrollment of patients will be temporary interrupted after the inclusion of first 6 patients in the trial. When 6 patients will complete the study treatment, a Safety Monitoring Committee will complete a safety evaluation.

The enrollment will then resume only if the study treatment combination is judged feasible and no major safety concerns arise.

The study primary endpoint will be the pathological complete response rate or pCR rate, defined as the percentage of patients, relative to the total of enrolled subjects in the intention-to-treat population, who will achieve a pathological complete response, as per central pathological review.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent.
2. Subjects must be 18 years old or older.
3. ECOG performance status of 0 to 1.
4. Histologically confirmed diagnosis of MCC amenable for radical surgery as defined by local or institutional surgical practices, based on multidisciplinary team assessment. Subjects must have one of the following stages of disease:

   1. Stage IIA - IIB- III (according to the AJCC staging system 8th edition)
   2. Local/Regional recurrent disease after primary surgery, as defined as total disease burden ≥ 1 cm diameter amenable for a radical intent surgery. Note: nodal disease without any known primary (in absence of a primary cutaneous site after a complete diagnostic/staging work-up including chest/abdomen CT-scan, dermatologic clinical examination and 18F-FDG-PET scan) can be enrolled and will be considered as Stage III.
5. Able to provide archival FFPE tumor samples (if collected within three months from study enrollment) or have a tumor amenable to pre-treatment biopsy. Excisional, incisional, or core- needle samples are acceptable. Fine needle aspirates are not allowed.
6. No prior systemic treatment or neoadjuvant radiation therapy.
7. Adequate bone marrow function characterized by the following at screening:

   1. Platelets ≥ 100 × 109/L
   2. Absolute neutrophil count (ANC) ≥1.5 x 109/L
   3. Hemoglobin ≥ 9.0 g/dL
8. Adequate renal function characterized by serum creatinine ≤ 1.5 × upper limit of normal (ULN) OR calculated by Cockroft-Gault formula or directly measured creatinine clearance ≥ 60 mL/min at screening for subject receiving cisplatin OR creatinine clearance ≥ 50 mL/min at screening for subject receiving carboplatin.
9. Adequate hepatic function characterized by the following at screening:

   1. Serum total bilirubin ≤ 1.5 × ULN and < 2 mg/dL. Note: Subjects with Serum total bilirubin ≥ 1.5 × ULN and conjugated bilirubin ≤ ULN or < 40% of total bilirubin are allowed.
   2. AST (SGOT) and/or ALT (SGPT) <2.5 x UNL.
10. Men must agree to take appropriate precautions to avoid fathering children (with at least 99% certainty) from screening through 6 months after the administration of study treatment and must refrain from donating sperm during this period. Permitted methods that are at least 99% effective in preventing pregnancy (see Appendix A) should be communicated to the participants and their understanding confirmed.
11. Women of childbearing potential must have a negative serum pregnancy test at screening and before the first dose on Day 1 and must agree to take appropriate precautions to avoid pregnancy (with at least 99% certainty) from screening through 180 days after the administration of any study drug. Permitted methods that are at least 99% effective in preventing pregnancy should be communicated to the participants and their understanding confirmed.
12. Women of non-childbearing potential (i.e. surgically sterile with a hysterectomy and/or bilateral oophorectomy OR ≥ 12 months of amenorrhea and at least 50 years of age) are eligible.
13. Willingness to comply with scheduled visits, treatment plan, laboratory tests and other study procedures.

Exclusion Criteria:

1. Prior systemic therapy for MCC, including chemotherapy and prior PD-1 or PD-L1-directed therapy.
2. Primary tumor or nodal metastasis fixed to the carotid artery, skull base or cervical spine.
3. Treatment with anticancer drugs, radiation therapy or participation in another interventional clinical study within 28 days before the first administration of study drug.
4. Distant metastases at any site.
5. Any known additional malignancy that is progressing or requires active treatment, or history of other malignancy within 2 years of study entry except for cured basal cell or squamous cell carcinoma of the skin, superficial bladder cancer, prostate intraepithelial neoplasm, carcinoma in situ of the cervix, or other noninvasive or indolent malignancy.
6. Impaired cardiovascular function or clinically significant cardiovascular diseases, including any of the following:

   1. History of acute myocardial infarction, acute coronary syndromes (including unstable angina, coronary artery bypass graft [CABG], coronary angioplasty or stenting) ≤ 6 months prior to start of study treatment;
   2. Symptomatic congestive heart failure (i.e., Grade 2 or higher), history or current evidence of clinically significant cardiac arrhythmia and/or conduction abnormality ≤ 6 months prior to start of study treatment, except atrial fibrillation and paroxysmal supraventricular tachycardia
7. History of autoimmune disease including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis.

   Note: Subjects with a history of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone may be eligible. Subjects with controlled type I diabetes mellitus on a stable insulin regimen, vitiligo or psoriasis not requiring systemic treatment may be eligible.
8. History of chronic conditions (i.e. COPD) requiring systemic immune-suppression in excess of physiologic maintenance doses of corticosteroids (> 10 mg of prednisone or equivalent).
9. Evidence of interstitial lung disease or active noninfectious pneumonitis.
10. History of organ transplant, including allogeneic stem cell transplantation.
11. History or current evidence of any condition, therapy or laboratory abnormality that might interfere with the subject's participation to the study or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
12. Know active hepatitis B [positive HBV surface antigen (HBsAg) result] or hepatitis C. Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA
13. Known uncontrolled HIV infection. HIV-positive patients are eligible if their CD4+ cell count amounts to 300 cells per μL or more; HIV viral load must be undetectable per standard of care assay, and they have to be compliant with antiretroviral treatment.
14. Active infections requiring systemic therapy, or systemic antibiotic use up to 10 days before Cycle 1 Day 1.
15. Live vaccines within 28 days prior to and for a duration of 90 days after the administration of study drug are forbidden.

    Note: Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, chickenpox/zoster, yellow fever, rabies, Bacillus Calmette Guérin, and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed. COVID-19 vaccine is allowed, with an interval of 2 days before and 2 days after the administration of study drugs;
16. Known hypersensitivity to platinum, etoposide or any of the excipients that cannot be controlled with standard measures (eg, antihistamines, corticosteroids).
17. Known allergy or hypersensitivity to any component of the study drug formulation.
18. Subjects who lack the ability or are unlikely, in the opinion of the investigator, to comply with the Protocol requirements.
19. Subjects who are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-12-07 (Actual); Primary Completion 2025-11-15 (Actual); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response rate (pCR rate) | 5 weeks
  Percentage of patients, relative to the total of enrolled subjects in the intention-to-treat population, who will achieve a pathological complete response, as per central pathological review. Pathological complete response will be defined as the absence of residual viable invasive cancer on evaluation of the complete resected tumor specimen and all sampled regional lymph nodes.

SECONDARY OUTCOMES:
Safety of the preoperative chemo-immunotherapy study regimen | 5 weeks
  Incidence of adverse events (AEs)
Safety of the preoperative chemo-immunotherapy study regimen | 5 weeks
  Incidence of serious adverse events (SAEs)
Safety of the preoperative chemo-immunotherapy study regimen a | 5 weeks
  G3/4 Toxicity Rate defined as the percentage of patients, relative to the total of enrolled subjects, experiencing any specific adverse event of grade 3/4, according to NCI-CTCAE v5.0, during the short-course preoperative chemo-immunotherapy study regimen
Safety of the preoperative chemo-immunotherapy study regimen a | 5 weeks
  Rate of surgery delay, defined as the proportion of patients receiving the short- course preoperative chemo-immunotherapy study regimen with surgery delayed > 4 weeks from the planned date due to a drug-related AE
Safety of the preoperative chemo-immunotherapy study regimen a | 5 weeks
  Surgical mortality
Patients' quality of life | 5 weeks
  Quality of life will be assessed through Patient reported outcomes (PRO) instrument: FACT-M Questionnaire
Impact of the short-course preoperative chemo-immunotherapy study regimen on patients' quality of life | 5 weeks
  Quality of life will be assessed through Patient reported outcomes (PRO) instrument: EQ-5D-5L
Relapse Free Survival | 24 months
  Relapse Free Survival will be defined as the time from enrollment to the first documentation of disease recurrence or death due to any cause, whichever occurs first.
Overall Survival | 24 months
  Overall survival will be defined as the time from enrollment to the date of death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Federica Morano, MD, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Locations (1):
- Fondazione IRCCS Istituto Nazionale dei Tumori di Milano, Milan, Italy

IPD SHARING:
Plan to Share IPD: No
The trial results concerning the primary, secondary and exploratory outcomes will be published according to the standard guidelines. IPD could eventually be requested to the Sponsor and Principal Investigator, who will carefully evaluate the formal and motivated request.

REFERENCES:
- [Background] Fields RC, Busam KJ, Chou JF, Panageas KS, Pulitzer MP, Allen PJ, Kraus DH, Brady MS, Coit DG. Recurrence after complete resection and selective use of adjuvant therapy for stage I through III Merkel cell carcinoma. Cancer. 2012 Jul 1;118(13):3311-20. doi: 10.1002/cncr.26626. Epub 2011 Nov 9. PMID 22072529
- [Background] D'Angelo SP, Bhatia S, Brohl AS, Hamid O, Mehnert JM, Terheyden P, Shih KC, Brownell I, Lebbe C, Lewis KD, Linette GP, Milella M, Georges S, Shah P, Ellers-Lenz B, Bajars M, Guzel G, Nghiem PT. Avelumab in patients with previously treated metastatic Merkel cell carcinoma: long-term data and biomarker analyses from the single-arm phase 2 JAVELIN Merkel 200 trial. J Immunother Cancer. 2020 May;8(1):e000674. doi: 10.1136/jitc-2020-000674. PMID 32414862
- [Background] Hodgson NC. Merkel cell carcinoma: changing incidence trends. J Surg Oncol. 2005 Jan 1;89(1):1-4. doi: 10.1002/jso.20167. PMID 15611998
- [Background] Heath M, Jaimes N, Lemos B, Mostaghimi A, Wang LC, Penas PF, Nghiem P. Clinical characteristics of Merkel cell carcinoma at diagnosis in 195 patients: the AEIOU features. J Am Acad Dermatol. 2008 Mar;58(3):375-81. doi: 10.1016/j.jaad.2007.11.020. PMID 18280333
- [Background] Harms KL, Healy MA, Nghiem P, Sober AJ, Johnson TM, Bichakjian CK, Wong SL. Analysis of Prognostic Factors from 9387 Merkel Cell Carcinoma Cases Forms the Basis for the New 8th Edition AJCC Staging System. Ann Surg Oncol. 2016 Oct;23(11):3564-3571. doi: 10.1245/s10434-016-5266-4. Epub 2016 May 19. PMID 27198511
- [Background] Becker JC. Merkel cell carcinoma. Ann Oncol. 2010 Oct;21 Suppl 7:vii81-5. doi: 10.1093/annonc/mdq366. PMID 20943647
- [Background] Chalabi M, Fanchi LF, Dijkstra KK, Van den Berg JG, Aalbers AG, Sikorska K, Lopez-Yurda M, Grootscholten C, Beets GL, Snaebjornsson P, Maas M, Mertz M, Veninga V, Bounova G, Broeks A, Beets-Tan RG, de Wijkerslooth TR, van Lent AU, Marsman HA, Nuijten E, Kok NF, Kuiper M, Verbeek WH, Kok M, Van Leerdam ME, Schumacher TN, Voest EE, Haanen JB. Neoadjuvant immunotherapy leads to pathological responses in MMR-proficient and MMR-deficient early-stage colon cancers. Nat Med. 2020 Apr;26(4):566-576. doi: 10.1038/s41591-020-0805-8. Epub 2020 Apr 6. PMID 32251400
- [Background] Topalian SL, Bhatia S, Amin A, Kudchadkar RR, Sharfman WH, Lebbe C, Delord JP, Dunn LA, Shinohara MM, Kulikauskas R, Chung CH, Martens UM, Ferris RL, Stein JE, Engle EL, Devriese LA, Lao CD, Gu J, Li B, Chen T, Barrows A, Horvath A, Taube JM, Nghiem P. Neoadjuvant Nivolumab for Patients With Resectable Merkel Cell Carcinoma in the CheckMate 358 Trial. J Clin Oncol. 2020 Aug 1;38(22):2476-2487. doi: 10.1200/JCO.20.00201. Epub 2020 Apr 23. PMID 32324435
- [Background] Gotwals P, Cameron S, Cipolletta D, Cremasco V, Crystal A, Hewes B, Mueller B, Quaratino S, Sabatos-Peyton C, Petruzzelli L, Engelman JA, Dranoff G. Prospects for combining targeted and conventional cancer therapy with immunotherapy. Nat Rev Cancer. 2017 May;17(5):286-301. doi: 10.1038/nrc.2017.17. Epub 2017 Mar 24. PMID 28338065